16.1.9 Documentation of Statistical Methods

# **Electronic Signature Page**



Document title: Statistical Analysis Plan

Sign-off status: FINAL

Digitally signed by:



| NAME, POSITION | ROLE | DATE TIME STAMP |
|---|---|---|
| | originator | 15-OCT-2021<br>22:39 (GMT+03:00) |
| | reviewer | 15-OCT-2021<br>22:41 (GMT +03:00) |
| | reviewer | 16-OCT-2021<br>10:56 (GMT +03:00) |
| COP ON | reviewer | 18-OCT-2021<br>10:28 (GMT +03:00) |
| BLC SUPPOS | approver | 18-OCT-2021<br>20:22 (GMT +03:00) |
| PUP dio silo | approver | 19-OCT-2021<br>15:45 (GMT+03:00) |
| PUBLIC SUPPORTS PUBLIC | | |
| This signoff page has been automatically generated to capture the digi | tal signatures of author | rized signatories. |

This signoff page has been automatically generated to capture the digital signatures of authorized signatories. Each record has been time-stamped and verified as authentic by certified software, providing evidence that the signed document has not been altered or tampered with post-signature.

Review Status: Final Version: 2.0 Version Date: 15OCT2021

# Ra Pharmaceuticals Inc (now part of UCB)

A MULTICENTER, OPEN-LABEL, UNCONTROLLED, STUDY OF RA101495 IN SUBJECTS WITH PAROXYSMAI LOBINURIA WHO HAVE COMPLETED A RA101495 EXTENSION STUDY OF RA101495 IN SUBJECTS WITH PAROXYSMAL NOCTURNAL HEMOGLOBINURIA WHO HAVE COMPLETED A RA101495 CLINICAL STUDY

RA101495-01.202 (UCB study PNH001) Protocol code:

This document cannot be used any externation and externation and exter **SAP Version:** Final 2.0

Review Status: Final

Version: 2.0

Version Date: 15OCT2021

# **DOCUMENT HISTORY**

# **VERSION HISTORY**

| Version # | Version Date |
|-----------|---------------|
| Final 1.0 | 09 April 2021 |
| Final 2.0 | 15OCT2021 |

# **REVISION HISTORY**

| Version # | Chapter | Revision Summary | Reason(s) for Revision |
|---|---|---|---|
| 1.0 | N/A | Initial release | N/A |
| 2.0 | 2 | CRF version updated | New CRF version |
| | 9.4 | Reason for treatment discontinuation removed from disposition summary | No separate treatment discontinuation reason was collected in addition to study discontinuation reason |
| | 9.6.4 | WHODrug version updated | Newer version used |
| | 9.8.3 | AE summary extended | Due to reporting requirements |
| | 9.11 | Clarification that no interim analysis was performed | No interim analysis was performed |
| | 10 | No analysis of CH50 | No data available |
| ocumer | Plication | nalysis was performed No analysis of CH50 | |


# **APPROVAL SIGNATURES**

| | STUDY TITI | <b>LE</b> : A MULTICENTER, OPEN-LABEL, U | NCONTROLLED, |
|---|---|---|---|
| | | N STUDY OF RA101495 IN SUBJECTS<br>AL HEMOGLOBINURIA WHO HAVE CO | MPLETED A RA101495 CLINICAL |
| | PROTOCOL | L <b>NUMBER:</b> RA101495-01.202 (UCB stu | udy PNH001) |
| | SAP Final 2 | .015OCT2021 | |
| | PSI<br>Author: | | Date: |
| | Signature: | | Date: |
| | Signature: | | Date: |
| | | | of Jo |
| | Signature: | JP 10 Silver | Date: |
| | Signature: | 15, 6 | Date: |
| | <u>UCB</u> | | |
| | Signature: | | Date: |
| | Signature | | Date: |
| 1/1/1/2 | | | |


# **TABLE OF CONTENTS**

| 1. | LIST | OF ABBREVIATIONS | 6 |
|---|---|---|---|
| 2. | INTR | ODUCTION | 8 |
| 3. | STUD | DY OBJECTIVES | 8 |
| | 3.1 | Objectives | 8 |
| 4. | STUD | DY DESCRIPTION | 8 |
| | 4.1 | Study Design | .O.8 |
| | 4.2 | Study Treatment | . 8 |
| | 4.3 | | |
| 5. | SAMI | Data and Safety Monitoring Board (DSMB) | و |
| 6. | ANAL | YSIS ENDPOINTS | <u>,</u> 9 |
| | 6.1 | Efficacy Endpoints | 9 |
| | 6.2 | Safety Endpoints | 9 |
| | 6.3 | Exploratory Endpoints | 9 |
| | 6.4 | Pharmacokinetic Endpoints | 9 |
| | 6.5 | Pharmacodynamic Endpoints | 9 |
| 7. | ANAL | YSIS POPULATIONS | 10 |
| 8. | СОНО | ORTS | 10 |
| 9. | ANAI | VTICAL DI AN AND STATISTICAL METHODS | 10 |
| ۶. | 9.1 | General Conventions and Statistical Considerations | 10 |
| | 9.2 | Definition of Reseline Study Visits and Visit Windows | 11 |
| | 9.3 | Handling of Missing Data | 17 |
| | 9.4 | Subject Disposition | 17 |
| | 9.5 | Definition of Baseline, Study Visits, and Visit Windows Handling of Missing Data | 12 |
| | 9.6 | Subject Characteristics | 13 |
| | 5.0 | 9.6.1 Baseline and Demographic Characteristics | 13 |
| | | 9.6.2 Medical History | 13 |
| | | 9.6.3 PNH Disease And Treatment History | 13<br>13 |
| | 9.7 | Efficacy Endpoints and Analysis | |
| | • | 9.7.1 Analysis of Efficacy Endpoints | 14 |
| | 9.8 | Safety Endpoints and Analysis | |
| | | 9.8.1 Exposure to Study Treatment | 14 |
| | | 9.8.2 Clinical Laboratory Evaluation | |
| | | 9.8.4 Immunogenicity | 21 |
| | | 9.8.5 Electrocardiogram | |
| | 00 ( | 9.8.6 Vital Signs and Other Safety Parameters | |
| | 9.9 | Exploratory Endpoints | |
| | | 9.9.2 FACIT-Fatigue | 25 |
| | <b>)</b> | 9.9.3 Mechanistic Biomarkers | 26 |
| O | 9.10 | | |
| <b>J</b> | | 9.10.1 Pharmacokinetics | |
| | 9.11 | Interim Analysis | |
| 10. | DFVT | ATIONS FROM ANALYSIS AS DESCRIBED IN THE PROTOCOL | |
| 11. | | GRAMMING SPECIFICATIONS | 29 |

| Stati | stical Analysis Plan: RA101495-01.202 / PNH001 | Review Status: Final Version: 2.0 |
|---|---|---|
| 12. | REFERENCES | 30 |
| 13. | APPENDIX I: LIST OF TABLES, LISTINGS, AND FIGURES | 31 |
| 14. | APPENDIX II. SCHEDULE OF ASSESSMENTS | 37 |
| | | :1'0 |
| | | Olli |
| | | .,0,0 |
| | | Sill NO. |
| | | S |
| | | ONS |
| | A A A | |
| | R all all a | |
| | CO. K. 1.0 | |
| | 1/2,000 5/0, | |
| | Po Air ans | |
| | Les to | |
| | 9,0 | |
| | Co. Co. | |
| | ~ (C) | |
| | Ull all of the | |
| 20 | | |
| .60 | | |
| Mis | | |
| | REFERENCES APPENDIX I: LIST OF TABLES, LISTINGS, AND FIGURES. APPENDIX II. SCHEDULE OF ASSESSMENTS CONFIDENTAL | |
| | CONFIDENTAL | |
| | . age <b>c</b> s. <b>c</b> . | |


# 1. LIST OF ABBREVIATIONS

| Abbroviotion | Full Torm |
|---|---|
| Abbreviation | Full Term Anti-drug Antibody Adverse Event Alkaline Phosphatase Alanine Aminotransferase |
| ADA | Anti-drug Antibody |
| AE | Adverse Event |
| ALP | Alkaline Phosphatase |
| ALT A DTT | Alanine Aminotransferase |
| aPTT/APTT | Activated Partial Thromboplastin Time |
| AST | Aspartate Aminotransferase |
| AUC | Area Under the Drug Concentration-time Curve |
| BMI | Body Mass Index |
| BUN | Blood Urea Nitrogen |
| C5 | Complement Component 5 |
| CH50 | Complement Total |
| cm | Centimeter |
| C <sub>max</sub> | Maximum Plasma Concentration |
| CPK | Creatine Phosphokinase |
| CRP | C-reactive Protein |
| CSR | Clinical Study Report |
| CTCAE | Common Terminology Criteria for Adverse Events |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| ELISA | Enzyme-linked Immunosorbent Assay |
| EQ-5D | EuroQol 5D Questionnaire |
| EORTC-QLQ-C30 | European Organization for Research and Treatment |
| | of Cancer-Quality of Life Questionnaire |
| FACIT-F | Functional Assessment of Chronic Illness Therapy- |
| | Fatigue Scale |
| GGT | Gamma-glutamyl Transferase |
| HR | Heart Rate |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonization |
| INR | International Normalized Ratio |
| ISR O | Injection Site Reaction |
| kg | Kilogram |
| LDH | Lactate Dehydrogenase |
| MAVE | Major Adverse Vascular event |
| MCH | Mean Corpuscular Hemoglobin |
| MCHC | Mean Corpuscular Hemoglobin Concentration |
| MCV | Mean Corpuscular Volume |
| MDRD | Modification of Diet in Renal Disease |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | Milligram |
| NČI | National Cancer Institute |
| PD | Pharmacodynamics |


| DIV Disamonda Lima Pian | l |
|---|---|
| PK Pharmacokinetics | l. |
| PNH Paroxysmal Nocturnal Hemoglobinuria | |
| PT Prothrombin Time PT Preferred Term PTT Partial Thromboplastin Time QOL Quality of Life RBC Red Blood Cell | |
| PT Preferred Term | |
| PTT Partial Thromboplastin Time | |
| QOL Quality of Life | |
| RBC Red Blood Cell | |
| SAE Serious Adverse Event | |
| SAP Statistical Analysis Plan | |
| SOC System Organ Class | |
| sRBC Sheep Red Blood Cell | |
| TEAE Treatment-emergent Adverse Event | |
| t Time to Corresponding Chay | |
| ULN Upper Limit of Normal | |
| VAS Visual Analogue Scale | |
| WBC White Blood Cell | |
| SLLOQ Below the Lower Limit of Quantification | |
| U.N. Upper Limit of Normal VAS Visual Analogue Scale WBC White Blood Cell <a href="https://doi.org/10.1001/j.j.com/bio/scale/">LLOQ</a> Below the Lower Limit of Quantification CONFIDENTAL | |
| CONFIDENTAL | |


## 2. INTRODUCTION

This statistical analysis plan (SAP) covers the analysis and reporting for protocol RA101495-01.202 dated 20 October 2016 and electronic case report form (eCRF) version 44 dated 22 March 2021. The following country-specific amendments are also reflected:

USA: Study Protocol amendment (version 03-FEB-2017)

Germany: Study Protocol amendment (version 03-MAY-2017)

Finland: Study Protocol amendment (version 24-FEB-2017)

UK: Study Protocol amendment (version 07-FEB-2017)

Denmark: Study Protocol amendment (version 11-APR-2017)

# 3. STUDY OBJECTIVES

## 3.1 **OBJECTIVES**

- have com all ben? To provide access to RA101495 for subjects with PNH who have completed a Ra Pharmaceuticals sponsored study, have demonstrated clinical benefit, and who wish to continue receiving RA101495 for treatment of PNH
- To evaluate the long-term safety and tolerability of RA101495 administered to subjects with PNH who have completed a Ra Pharmaceuticals sponsored RA101495 clinical study
- To evaluate the long-term preliminary efficacy of RA101495 administered to subjects with PNH who have completed a Ra Pharmaceuticals sponsored RA101495 clinical study
- To obtain periodic PK and PD data to confirm long-term maintenance of steady-state RA101495 plasma levels and sustained inhibition of hemolysis and complement

# 4. STUDY DESCRIPTION

## 4.1 STUDY DESIGN

The design is a multicenter, open-label, extension study for subjects with PNH who have successfully completed a qualifying Ra Pharmaceuticals sponsored RA101495 (zilucoplan) clinical study (RA101495-01.201 or RA101495-01.203). Subjects will continue to receive the final maintenance dose they were receiving in the qualifying study, as long as safety, tolerability, PK and PD data (from the qualifying study or this extension study) continue to demonstrate benefit. If additional data support a change in dose level for an individual subject in this extension study, investigators may increase or decrease the maintenance dose level, based on safety and PD findings, and in consultation with the medical monitor. All subjects will continue to be followed carefully for any evidence of meningococcal and/or other infection.

### 4.2 STUDY TREATMENT

All eligible subjects will receive open-label RA101495 daily by SC self-injection. The starting


dose in the extension study will be the same as the final maintenance dose the subject was receiving in the qualifying study. The IMP (RA101495) will continue to be provided by the sponsor until RA101495 is approved and available in the territory or the sponsor terminates development of RA101495 for PNH.

# 4.3 DATA AND SAFETY MONITORING BOARD (DSMB)

No DSMBs are scheduled for this study.

# 5. SAMPLE SIZE AND POWER CALCULATION

Sample size will be determined by the number of eligible subjects completing a qualifying RA101495 clinical study. No formal statistical sample size estimates were performed.

# 6. ANALYSIS ENDPOINTS

# 6.1 EFFICACY ENDPOINTS

Serum LDH levels, total bilirubin, total hemoglobin, free hemoglobin, haptoglobin, reticulocytes, and hemoglobinuria, at each of the scheduled assessment time-points.

# 6.2 SAFETY ENDPOINTS

Safety assessments will include an evaluation of AEs and SAEs (including major adverse vascular event (MAVE criteria)), clinical laboratory tests, ECGs, vital signs, and physical examinations.

# 6.3 EXPLORATORY ENDPOINTS

- Quality of life (QOL) questionnaires (e.g. EORTC QLQ-C30 and FACIT-Fatigue)
- Mechanistic biomarkers (e.g. complement function, complement proteins, biomarkers of inflammation, biomarkers for thrombosis, biomarkers of liver function) to be summarized in a separate report.

# 6.4 PHARMACOKINETIC ENDPOINTS

Plasma concentrations of RA101495 and its major metabolite(s)

# 6.5 PHARMACODYNAMIC ENDPOINTS

- CH<sub>50</sub>
- Sheep RBC (sRBC) lysis for the classical complement pathway
- Wieslab ELISA for alternative complement pathway
- C5 levels

Note: CH<sub>50</sub> is not analyzed as it is not collected.


# 7. ANALYSIS POPULATIONS

# **SAFETY POPULATION**

The Safety Population will include all subjects who receive at least 1 injection of RA101495 on or after Day 1 of this extension study (RA101495-01.202).

# PHARMACOKINETIC POPULATION

The PK population will include all subjects in the safety Population who have at least 1 plasma sample obtained for PK assessment.

# PHARMACODYNAMIC POPULATION

The PD population will include all subjects in the safety Population who have at least 1 plasma sample obtained for PD assessment.

# 8. COHORTS

The following cohorts of the study populations will be used for analyses

# **Eculizumab Naïve Subjects**

This will include all subjects who have not received eculizumab for treatment of PNH (i.e., subjects from study RA101495-01.201 Cohort A (Naïve)).

# **Eculizumab Switch Subjects**

This will include all subjects who have received treatment with eculizumab for at least 6 months prior to Screening. (i.e., subjects from study RA101495-01.201 Cohort B (Switch)).

# Inadequate Response to Eculizumab Subjects

This will be a subset of the Eculizumab Switch Subjects coming from the RA101495-01.203 study, including all subjects who had an inadequate response to eculizumab defined as having received eculizumab for at least 6 months plus meeting one or both of the following criteria:

- A documented lactate dehydrogenase (LDH) level ≥ 1.5 x the upper limit of normal (ULN) within 90 days prior to Screening
- Presence of a known C5 mutation conferring resistance to eculizumab.

# 9. ANALYTICAL PLAN AND STATISTICAL METHODS

# 9.1 GENERAL CONVENTIONS AND STATISTICAL CONSIDERATIONS

Data will be summarized by eculizumab-naïve, eculizumab switch, and inadequate responder groups with all doses within these groups being pooled.


version Date: 150C12021

All clinical study data will be presented in Subject data listings. Descriptive statistics (n, mean, standard error of the mean, standard deviation, median, minimum, and maximum) will be calculated by cohort for continuous variables.

Counts and proportions will be presented by cohort for categorical and ordinal variables. If there are missing values, the number of missing values will be presented, but without a percentage and the number of non-missing values used as the denominator.

Means, medians, standard deviations, standard error of the mean, and confidence intervals will be reported to one decimal place more than the data reported on the CRF or by the laboratory/vendor. Minimum and maximum will be reported to the same number of decimal places displayed on the CRF or by the laboratory/vendor.

Assuming that an endpoint is expected to be in a numeric format, all non-numeric values entered as "< X.XX" or "> Y.YY" will be analyzed as X.XX or Y.YY, respectively.

# 9.2 DEFINITION OF BASELINE, STUDY VISITS, AND VISIT WINDOWS

Unless otherwise specified, a subject's baseline will be the value from the Screening/Day 1 value of this study. The Screening Visit will generally coincide with the qualifying study end of study visit. Should the last qualifying study visit be missing, the last available observation in the qualifying study will be used. All screening assessments are expected to be the same as those for the end of qualifying study visit and do not need to be repeated unless clinically indicated. Change from baseline will be calculated by subtracting the baseline value from the post-dose assessment for each subject (i.e. post-dose – baseline). Percent change from baseline will be calculated as 100×change score/ baseline score.

There will be no windowing of study visits in this study. However, the following rules will be used to assign display values of study visits:

| Visit in SDTM | Display in Analysis | Comment |
|---------------|---------------------|------------------------|
| | Baseline | Assigned per SAP above |
| Day 30 | Month 1 | |
| Day 60 | Month 2 | |
| Day 90 | Month 3 | |
| Day 120 | Month 4 | |
| Day 150 | Month 5 | |
| Day 180 | Month 6 | |
| Day 210 | Month 7 | |
| Day 240 | Month 8 | |
| Day 270 | Month 9 | |
| Day 300 | Month 10 | |


| Day 330 | Month 11 |
|---|---|
| Day 360 | Month 12 |
| Day 390 | Month 13 |
| Day 420 | Month 13 Month 14 Month 15 Month 16 |
| 3 Month Visit 1 | Month 15 |
| 3 Month Visit 1-1 | Month 16 |
| 3 Month Visit 1-2 | Month 17 |
| 3 Month Visit 2 | Month 18 |
| 3 Month Visit 2-1 | Month 19 |
| 3 Month Visit 2-2 | Month 20 |
| | 10, 10 |
| 3 Month Visit x | Add one month from previous |
| 3 Month Visit x-1 | Add one month from previous |
| 3 Month Visit x-2 | Add one month from previous |
| 3 Month Visit 12 | Month 50 |
| 3 Month Visit 12-1 | Month 51 |
| 3 Month Visit 12-2 | Month 52 |
| Final Study Visit | Final Study Visit Combine all subjects' last visit as reported in CRF regardless of study duration. |

# 9.3 HANDLING OF MISSING DATA

Unless otherwise stated, missing data will not be imputed; observed cases will be used in the analyses.

# 9.4 SUBJECT DISPOSITION

A disposition of all consented subjects will be provided. This will include a breakdown of subjects who consented, were treated, and were discontinued from the study. The primary reason for discontinuation from the study will be summarized. Additionally, a summary of subjects included in the analysis populations outlined in Section 7 will be included.

Listings of all the disposition data, including date of IC signed, date and reason of discontinuation, and protocol version will be created.

# 9.5 PROTOCOL DEVIATIONS

Major Protocol deviations will be summarized. Protocol deviations will be presented in a listing that will include all deviations that lead to a subject being withdrawn from the per-protocol population.


# 9.6 SUBJECT CHARACTERISTICS

# 9.6.1 BASELINE AND DEMOGRAPHIC CHARACTERISTICS

Subject demographics and baseline characteristics will be summarized for the safety population.

Descriptive statistics will be provided for age, height, weight, and body mass index (BMI, calculated as weight in kilograms divided by height in meters squared). Frequencies and percentages will be tabulated for sex, race, ethnicity, and country.

Age will be calculated as (informed consent date in the RA10495-01.202 study – date of birth + 1)/365.25, truncated and displayed as years. Should either or both the month and day of birth be missing, the date will be set to June 1<sup>st</sup>.

BMI will be calculated as weight (kg)/height<sup>2</sup> (m<sup>2</sup>), using the weight and height measurements obtained at screening.

Inches will be converted to centimeters with 2.54 cm being equal to 1 in

# 9.6.2 MEDICAL HISTORY

Medical history will be summarized with data that was collected at the screening visit of the subject's qualifying study will be coded using MedDRA version 19.1 or higher. The summary in this section will be run for the safety Population. The number of Subjects with prior and concurrent conditions by preferred term will be output.

# 9.6.3 PNH DISEASE AND TREATMENT HISTORY

Separate listings for PNH disease history and PNH treatment will be created.

# 9.6.4 PRIOR AND CONCOMITANT MEDICATIONS

All concomitant medications ongoing from the qualifying study will be documented. All medications will be documented using WHODrug Global Format B3 September 2020 or higher. Concomitant medications include any prescription or over-the-counter medication that is ongoing on Day 1 or that is initiated following the first dose of study drug on Day 1. A medication will be classified as a prior medication if its start date is earlier than the date of first study drug administration and is not ongoing at the first dose.

Incidence of prior and concomitant medications will be presented by therapeutic area, and preferred (generic) drug name for the safety population


### 9.7 **EFFICACY ENDPOINTS AND ANALYSIS**

# 9.7.1 ANALYSIS OF EFFICACY ENDPOINTS

Efficacy endpoints will be summarized at each scheduled assessment time point using descriptive statistics for the observed and change from baseline values for safety population.

Efficacy assessments include:

# 9.8

Safety analysis results will be presented using the safety Population.

# 9.8.1

y population.

Reticulocytes

Hemoglobinuria using a urine colorimetric system.

SAFETY ENDPOINTS AND ANALYSIS

nalysis results will be presented using the safety Por

EXPOSURE TO STUDY TREATMENT

ere required to self administer P roroximately the same time
the qualifying study is ted. On days or red after is Subjects were required to self administer RA101495 as a SC injection once daily (every 24 hours at approximately the same time each day). On Day 1, the last dose administered on the final day of the qualifying study was considered the first dose on the extension study and was not be repeated. On days of the scheduled study visit at the investigator site, the dose was to be administered after the blood work was completed at the investigator site

Dose-levels will be summarized from the start of this study. The number of subjects with an increase in dose and decrease in dose (relative to the dose at the start of the study) will be summarized.

# 9.8.2 CLINICAL LABORATORY EVALUATION

Data listings will be produced for all collected laboratory data including hematology, chemistry, and coagulation and urinalysis. Laboratory values outside laboratory's normal ranges will be flagged as H (high, above normal) or L (low, below normal) in laboratory data listings.

# (A) CLINICAL CHEMISTRY, HEMATOLOGY, AND COAGULATION ANALYTES

Hematology, Serum Chemistry, Coagulation, C-reactive protein, and Creatine phosphokinase analyte, and Liver Function Test (see Table 3) values and change from baseline will be tabulated using descriptive statistics at each planned visit. The data will be presented in separate listings.

Review Status: Final Version: 2.0


Table 3: Clinical Chemistry, Hematology, and Coagulation Analytes

| Clinical Chemistry | Hematology |
|---|---|
| alanine aminotransferase (ALT) | |
| albumin | :49 |
| alkaline phosphatase (ALP) | hematocrit |
| amylase | hematocrit hemoglobin mean corpuscular hemoglobin (MCH) mean corpuscular hemoglobin concentration (MCHC) mean corpuscular volume (MCV) platelet count RBC count white blood cell (WBC) count and differential (%) |
| aspartate aminotransferase (AST) | mean corpuscular hemoglobin (MCH) |
| bicarbonate | mean corpuscular hemoglobin concentration |
| bile acids | (MCHC) |
| bilirubin (direct, and indirect) | (MCIC) |
| blood urea nitrogen (BUN) | mean corpuscular volume (MCV) |
| calcium | platelet count |
| chloride | RBC count |
| creatinine | |
| gamma-glutamyl transferase (GGT) | white blood cell (WBC) count and differential (%) |
| glucose | Coagulation |
| lipase | international normalized ratio (INR)/prothrombin time |
| potassium | (PT) |
| sodium | fibrinogen partial thromboplastin time (PTT) or activated |
| total protein | partial thromboplastin time (aPTT or APTT) |
| uric acid | Other |
| 10° 00' | C-reactive protein (CRP) |
| 20, 20, 0 | creatine phosphokinase (CPK) |

# (B) URINALYSIS

Urinalysis will be performed for measurement of pH, specific gravity, protein (qualitative), glucose (qualitative), ketones (qualitative), bilirubin (qualitative), urobilinogen, occult blood, hemoglobin, and cells.

Urinalysis values will be tabulated using descriptive statistics at each planned visit.

# (C) PREGNANCY TEST

A urine dipstick pregnancy test (human chorionic gonadotropin) will be performed on female subjects of childbearing potential. These results will be listed.

# (D) PNH CLONE

PNH clone size will be determined by peripheral blood flow cytometry analysis (RBCs and **CONFIDENTAL** 

Review Status: Final Version: 2.0


granulocytes) and is performed every 3 months. These results will be summarized and listed.

### 9.8.3 **ADVERSE EVENTS**

Adverse events will be coded using MedDRA (version 19.1 or higher). All events will be summarized and presented by Incidence rates for treatment-emergent adverse events (TEAEs by maximum severity and SAEs will be summarized. These summaries will be provided regardless of causality and for events that are considered possibly related to treatment with RA101495.

TEAEs are defined as follows:

- An AE that occurs after a subject's initial treatment RA101495 start for this study (RA101495-01.202) that was not present at the time of treatment start; or
- An AE that increases in severity after treatment start in this study, if the event was present at the time of treatment start.

TEAEs will be summarized for each cohort.

AEs occurring before the first dose of study drug in this study will be summarized separately and included in the overall AE analysis as appropriate.

The following TEAE summaries will be provided and, where applicable, summarized by system organ class, and preferred term:

- Overall summary of Treatment Emergent Adverse Events
- Incidence of Treatment Emergent Adverse Events
- Incidence of Non-serious Treatment Emergent Adverse Events
- Incidence of Treatment Emergent Adverse Events by Maximum Severity
- Incidence of Treatment Emergent Adverse Events by Relationship to Study Drug
- Incidence of Treatment Emergent Adverse Events Leading to Study Discontinuation
- Incidence of Serious Treatment Emergent Adverse Events.
- Incidence of Treatment Emergent Adverse Events above Reporting Frequency Threshold of 5%
- Incidence of Non-Serious Treatment Emergent Adverse Events above Reporting Frequency Threshold of 5%


- Incidence of TEAEs Leading to Death
- Incidence of treatment-related TEAEs Leading to Death\*
- Incidence of treatment-related serious TEAEs \*
- Incidence of treatment-related TEAEs leading to study drug discontinuation\*
- Incidence of Grade 3 or greater TEAEs\*
- Incidence of treatment-related Grade 3 or greater TEAEs\*

(\*: only in overall summary)

d at least c For these summaries, the number and percentage of subjects who experienced at least one of the TEAE as well as (where applicable) the number and percentage of subjects who experienced each specific SOC and PT will be presented. The corresponding number of TEAEs will also be presented, where applicable.

For the presentation of TEAE incidences, the SOCs will be sorted alphabetically, and within SOC, the preferred term (PT) will be used and presented by decreasing total frequency.

# (A) DETERMINING TREATMENT EMERGENT WITH ADVERSE EVENT DATES

The following rules apply when determining if an AE is treatment-emergent in the scenario where the start date is missing or partially missing. These rules provide an algorithm to "impute" a complete AE start date which will then be used to determine if the AE is treatment emergent.

# AE start date missing day and month

- If the year is the same as the year of the treatment start date, the day and month of the date of treatment start date will be assigned to the missing fields.
- If the year is prior to the year of the treatment start date, December 31 will be assigned to the missing fields.
- If the year is after the year of the date of the treatment start date, January 1 will be assigned to the missing fields.

# AE start date missing month only:

The day will be treated as missing, and both month and day will be replaced according to the above procedure.

# AE start date missing day only:

If the month and year are the same as the month and year of the treatment start date, the day of the treatment start date will be assigned to the missing day.


If either the year is before the year of the date of the treatment start date or if both years are the same but the month is before the month of the treatment start date, the last day of the month will be assigned to the missing day.

If either the year is after the year of the treatment start date or if both years are the same but the month is after the month of the treatment start date, the first day of the month will be assigned to the missing day.

# AE start date completely missing:

- If the AE end date is complete and after the treatment start date, the treatment start date will be assigned to the missing start date.
- If the end date is complete and before the treatment start date, the end date will be assigned to the missing start date
- Otherwise the AE start date will be assigned the treatment start date

If the end date is complete and the imputed start date as above is after the end date, the start date will be imputed by the end date.

# ADVERSE EVENTS OF SPECIAL INTEREST

(I) THROMBOTIC ADVERSE EVENTS

All be a will be ever and any extension and any A separate table for thrombotic TEAEs will be presented, summarizing TEAEs by SOC and PT. The events in Table 1 (Hillmen, 2007]) will be evaluated in the assessment of thrombotic

Review Status: Final Version: 2.0


Table 1: Thrombotic Event Description (MAVE Criteria)

| MAVE Criteria | AE Preferred Term Mapping | |
|---|---|---|
| Thrombophlebitis/Deep vein | Preferred Term: 10051055 Deep vein thrombosis | |
| thrombosis | Preferred Term: 10043570 Thrombophlebitis | |
| Pulmonary embolus | Preferred Term: 10037377 Pulmonary embolism | :4) |
| Myocardial infarction | Preferred Term: 10028596 Myocardial infarction | noi1 |
| Transient ischemic attack | Preferred Term: 10044390 Transient ischaemic attack | |
| Renal vein thrombosis | Preferred Term: 10038548 Renal vein thrombosis | · k. |
| Acute peripheral vascular occlusion | Preferred Term: 10053648 Vascular occlusion | 0, |
| Amputation (non-traumatic, non- | Preferred Term: 10061627 Amputation | |
| diabetic) | | ) |
| Mesenteric/Visceral vein thrombosis | Preferred Term: 10027402 Mesenteric vein thrombosis | |
| iviesemente/ v iscerar vein timoiniousis | Preferred Term: 10077829 Visceral venous thrombosis | |
| Unstable angina | Preferred Term: 10002388 Angina unstable | |
| Mesenteric/Visceral arterial | Preferred Term: 10027397 Mesenteric artery thrombosis | |
| thrombosis | Lower level term: 10043611 Thrombosis arterial | |
| Hepatic/Portal vein thrombosis | Preferred Term: 10019713 Hepatic vein thrombosis | |
| Trepatic/Tortal vein unombosis | Preferred Term: 10036206 Portal vein thrombosis | |
| Dermal thrombosis | Lower level term: 10042545 Superficial phlebothrombosis | |
| | Preferred Term: 10017711 Gangrene | |
| Gangrene (non-traumatic, non- | Preferred Term: 10009971 Colon gangrene | |
| diabetic) | Preferred Term: 10017954 Gastrointestinal gangrene | |
| Cerebral arterial | Preferred Term: 10008190 Cerebrovascular accident | |
| occlusion/cerebrovascular accident | Preferred Term: 10008089 Cerebral artery occlusion | |
| Cerebral venous occlusion | Preferred Term: 10076895 Cerebral vascular occlusion | |
| Renal arterial thrombosis | Preferred Term: 10038380 Renal artery thrombosis | |

Abbreviation: MAVE=major adverse vascular event.

# (II) HEPATIC ADVERSE EVENTS

Hepatic TEAEs and will be summarized separately by SOC, PT, and cohort. Liver function tests will be summarized by changes from baseline and graded in severity using the NCI CTCAE (Version 4.03) criteria.

These AEs will defined using MedDRA SMQs as:

Drug related hepatic disorders – comprehensive search (SMQ)(20000006) excluding liver neoplasms, malignant and unspecified (SMQ)(20000011) and liver neoplasms, benign (SMQ)(20000012).

# (III) PANCREATIC ENZYME ELEVATION

Pancreatic enzyme elevation will be reported as incidence of baseline and post baseline grades per NCI CTCAE (Version 4.03) criteria for increased amylase (Preferred Term "Amylase


- er and severity authorization severe)

  severe)

  severe)

  rate that the least to support and any attacher any

Review Status: Final Version: 2.0


**Table 2: Grading the Severity of Local Injection Site Reactions** 

| Local Reaction<br>to Injectable<br>Product | Grade 1<br>(Mild) | Grade 2<br>(Moderate) | Grade 3<br>(Severe) | Grade 4<br>(Potentially Life<br>Threatening) | :121 |
|---|---|---|---|---|---|
| Pain | Does not interfere with activity | Repeated use of<br>non-narcotic pain<br>reliever >24 hours or<br>interferes with<br>activity | Any use of narcotic pain reliever or prevents daily activity | Emergency room<br>visit or<br>hospitalization | ofile of |
| Tenderness | Mild discomfort<br>to touch | Discomfort with movement | Significant discomfort at rest | Emergency room visit or hospitalization | |
| Erythema/<br>redness | 2.5 to 5.0 cm | 5.1 to 10.0 cm | >10.0 cm | Necrosis or exfoliative dermatitis | |
| Induration/<br>swelling | 2.5 to 5.0 cm and does not interfere with activity | 5.1 to 10.0 cm or interferes with activity | >10.0 cm or prevents daily activity | Necrosis | |

The Injection site reactions CRF page has the date of assessment but is not specifically connected to a study visit (even though the assessment is planned to be done in conjunction with visits). Study visit will be assigned algorithmically based on the visit start and end dates and the actual ISR assessment date.

ISRs will be further analysed by SOC and PT for high level terms "injection site reactions", and "administration site reactions".

# (C) TEAE WITH SOC "INFECTIONS AND INFESTATIONS"

TEAEs related to infection will be summarized separately by system organ class, preferred term, and cohort. These are defined as those with "infections and infestations" as their system organ class.

# 9.8.4 JMMUNOGENICITY

No analysis of immunogenicity will be performed.

# 9.8.5 ELECTROCARDIOGRAM

Descriptive statistics for ECG parameters (i.e. heart rate (HR), PR interval, RR interval, QRS interval, QT interval, and QTcB intervals, and QTcF intervals) at each assessment timepoint will


be presented. The interpretation of ECG will be summarized at each visit.

QTc intervals will be calculated using both Fridericia's and Bazett's corrections, with the formulae:

Fridericia's correction: QTc = QT/RR<sup>0.33</sup>

Bazett's correction: QTc =QT/RR<sup>0.5</sup>.

# 9.8.6 VITAL SIGNS AND OTHER SAFETY PARAMETERS

Descriptive statistics for the actual value at each timepoint and the change from baseline to each post baseline timepoint in systolic and diastolic BP, heart rate, and body temperature will be tabulated by cohort and overall.

The complete set of physical examination findings will be provided in listings. Clinically significant physical examination abnormalities will be included and summarized as AEs if appropriate.

Grade 3 and 4 of increased lipase and amylase levels over baseline levels will be tabulated.

# 9.9 EXPLORATORY ENDPOINTS

All exploratory analyses will be done for the safety population.

# 9.9.1 EORTC QLQ-C30

Summary statistics for each scales/items scores will be presented as well as the corresponding change from baseline scores for each scheduled assessment time-point.

# Global health status

Global health status/Qol

# **Functional scales**

- Physical functioning
- Role functioning
- Emotional functioning
- Cognitive functioning
- Social functioning

# Symptom scales/items

Fatigue


- Nausea and vomiting
- Pain
- Dyspnoea
- Insomnia
- Appetite loss
- Constipation
- Diarrhoea
- Financial difficulties.

ed into 5 function (Table 4). The EORTC QLQ-C30 consists of 30 questions, which are incorporated into 5 functional domains (physical, role, cognitive, emotional, and social domains; see Table 4); a global health status/global QOL scale; 3 symptom scales (fatigue, pain, and nausea and vomiting scales); 6 single items that assess additional symptoms (e.g. dyspnea, appetite loss, sleep disturbance, constipation, and diarrhea); and the perceived financial burden of illness treatment (Aaronson, 1993; Aaronson, 1996). Subjects answer questions based on symptoms/status over the preceding week.

The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items.

Each of the multi-item scales includes a different set of items - no item occurs in more than one scale.

All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.

- a high score for a functional scale represents a high / healthy level of functioning
- a high score for the global health status / QoL represents a high QoL,
- a high score for a symptom scale / item represents a high level of symptomatology / problems.

The principle for scoring these scales is the same in all cases:

- 1. Estimate the average of the items that contribute to the scale; this is the raw score.
- 2. Use a linear transformation to standardize the raw score, so that scores range from 0 to 100; a higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.

CONFIDENTAL 


Table 4: Scoring the EORTC QLQ-C30

| Table 4. Scotting the LOKTO | <b>4_4</b> 00 | | | | |
|---|---|---|---|---|---|
| | Scale | Number of Items | Item<br>Range* | Item<br>Numbers | Functional scales |
| Global health status / QoL | | | | | |
| Global health status/QoL | QL2 | 2 | 6 | 29, 30 | |
| Functional scales | | | | | 0 |
| Physical functioning | PF2 | 5 | 3 | 1 to 5 | P) W |
| Role functioning | RF2 | 2 | 3 | 6, 7 | 5ns |
| Emotional functioning | EF | 4 | 3 | 21 to 24 | F |
| Cognitive functioning | CF | 2 | 30 | 20, 25 | F |
| Social functioning | SF | 3 5/1 | 3 5 | 26, 27 | F |
| Symptom scales / items | 200% | 10 | 5 | | |
| Fatigue | FAC | 30+ | 3 | 10, 12, 18 | |
| Nausea and vomiting | NV | 2 | 3 | 14, 15 | |
| Pain | PA | 2 | 3 | 9, 19 | |
| Dyspnoea Control Insomple | DY | 1 | 3 | 8 | |
| Insomnia | SL | 1 | 3 | 11 | |
| Appetite loss | AP | 1 | 3 | 13 | |
| Constipation | СО | 1 | 3 | 16 | |
| Diarrhoea | DI | 1 | 3 | 17 | |


| Financial difficulties | FI | 1 | 3 | 28 |
|------------------------|----|---|---|----|
|------------------------|----|---|---|----|

<sup>\*</sup> Item range is the difference between the possible maximum and the minimum response to individual items; most items take values from 1 to 4, giving range = 3. The exceptions are the items contributing to the global health status/QoL, which are 7-point questions with range = 6,

For all scales, the Raw Score is the mean of the component items.

For functional scales the score is:

Score = 
$$\{1 - (Raw score - 1)/(range)\} \times 100$$

and for Symptom scales/items and Global health status/QoL:

Score = 
$$\{(Raw score - 1)/(range)\} \times 100$$
.

Due to the potential for non-normal data, the change from baseline for the EORTC QLQ-C30 scales will be assessed by a two-sided Wilcoxon signed-rank test.

### 9.9.2 **FACIT-FATIGUE**

The overall FACIT-Fatigue score and the individual 13 item scores will be summarized as well as the corresponding change from baseline scores for each scheduled assessment time-point. Shift tables displaying the individual item values from baseline to each post-baseline visit will

Jue Scale is a 13-item, easy to admigue during their usual daily activities over ared on a five point ordinal scale (4 = not at all twebster, 2003].

The items and scoring algorithm are given in Table 5. The FACIT-Fatigue Scale is a 13-item, easy to administer tool that measures an individual's level of fatigue during their usual daily activities over the preceding week. The level of fatigue is measured on a five point ordinal scale (4 = not at all fatigued to 0 = very much fatigued)




# 9.9.3 MECHANISTIC BIOMARKERS

A separate analysis plan will be prepared for mechanistic biomarkers.

# 9.10 OTHER ENDPOINTS AND ANALYSIS

# 9.10.1 PHARMACOKINETICS

All following pharmacokinetic endpoints will be summarized using descriptive statistics.

• Plasma concentrations of RA101495 and its major metabolites

# 9.10.2 PHARMACODYNAMIC

Pharmacodynamic endpoints will be summarized at each scheduled assessment time point using descriptive statistics for the observed and change from baseline values.

Note: CH<sub>50</sub> is not analyzed as it is not collected.


This document cannot be used any extensions of variations the real and any extensions of variations are also as a variation of variations and variations of variations are also as a variation of variations of variations and variations of variations are also as a variation of variations of


# 10. DEVIATIONS FROM ANALYSIS AS DESCRIBED IN THE **PROTOCOL**

- 1. Due to the small number of subjects increasing doses, all analysis is done on the pooled cohorts instead of by dose level.
- 2. Due to some injections being done away from the clinic, total number of injections will not be summarized.
- 3. No analyses will be done on maximum plasma concentration, time to maximum concentration, or area under the drug-concentration time curves.
- 4. Due to the small number of subjects in the study, no analysis will be done on the perprotocol population. Similarly no hypothesis testing will be done on study endpoints.
- 5. Pancreatic enzyme elevation will not be summarized as AEs, but using the incidence of NCI CTCAE grades for amylase and lipase.
- 6. TEAEs for infections will not be restricted to Neisseria meningitidis
- will be performed.

  afformed.

  afformed.

  A politication and a politic 7. No analysis will be done on subject-years of exposure.
  - 8. No analysis of immunogenicity (ADA) will be performed

CONFIDENTAL 


### 11. PROGRAMMING SPECIFICATIONS

The margins should be at least 1.50 inches for the binding edge and 1.0 inches for all others.

In the top left portion of each table/listing, the protocol pure!

line a table/listing number 5." be displayed. Horizontal lines will appear after the column heading of the table/listing. Footnotes will be put under the main body of text at the bottom of the page. The SAS program name will appear bottom left in a string and the page number will appear on the bottom light corner of each table/listing. The date and time of creation of table/listing will appear bottom left under to the SAS program name line.

Jes and not manda , 07MAY2002 o given in section below.ck-Up (TFLs document. Courier New 8-point bold font will be used for all tables and listings. Usually, a landscape layout is suggested for both tables and listings, but it is not mandatory. Any date information in the listing will use the date9. format, for example, 07MAY2002 or other appropriate formats.

The list of tables, listings, and figures is given in section below. Shells for unique tables and


# 12. REFERENCES

Aaronson NK, Ahmedzai S, Bergman B, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst 1993;85:365-376.

Aaronson NK, Cull A, Kaasa S, et al. The European Organization for Research and Treatment of cologarials 2n.

.t of chronic illness to pretation. Health Qual La pretation. Health Qual La pretation and any angle of the Cancer (EORTC) modular approach to quality of life assessment in oncology: an update In: Spilker B, ed. Quality of Life and Pharmacoeconomics in Clinical Trials. 2nd Ed. New York,

Webster K, Cella D, and Yost K. The functional assessment of chronic illness therapy (FACIT) measurement system: properties, applications, and interpretation. Health Qual Life Outcomes

Review Status: Final


# APPENDIX I: LIST OF TABLES, LISTINGS, AND FIGURES ition All Enrolled Subjects Deviations Safety Population Treatment Safety Population Concurrent Conditions Safety Population afety Population DH Levels (U/L) Safety S 13.

Table 14.1.1.1 Subject Disposition All Enrolled Subjects

Table 14.1.1.2 Major Protocol Deviations Safety Population

Table 14.1.2 Subject Demographics and Baseline Characteristics Safety Population

Table 14.1.3 Exposure to Study Treatment Safety Population

Table 14.1.4 Medical History and Concurrent Conditions Safety Population

Table 14.1.5.1 Concomitant Medication Safety Population

Table 14.1.5.2 Prior Medication Safety Population

Table 14.2.1 Summary of Serum LDH Levels (U/L) Safety Population

Table 14.2.2 Summary of Total Bilirubin Values (umol/L) Safety Population

Table 14.2.3 Summary of Total Hemoglobin Values (g/L) Safety Population

Table 14.2.4 Summary of Free Hemoglobin Values (mg/dL) Safety Population

Table 14.2.5 Summary of Haptoglobin Values (g/L) Safety Population

**CONFIDENTAL** 

Review Status: Final


Table 14.2.6 Summary of Reticulocytes Values (10^12/L) Safety Population

Table 14.2.7 Summary of Hemoglobinuria Values Safety Population

Table 14.2.8 Summary of EORTC QLQ-C30 Safety Population

Table 14.2.9.1 Summary of FACIT-Fatigue: Overall Score Safety Population

Table 14.2.9.2 Summary of FACIT-Fatigue: Individual Items Safety Population

Table 14.2.9.3 Summary of FACIT-Fatigue: Items Shift Table Safety Population

Table 14.2.10 Summary of CH50 Values Pharmacodynamic Population

Table 14.2.11 Summary of sRBC Values Pharmacodynamic Population

Table 14.2.12 Summary of Wieslab ELISA Values Pharmacodynamic Population

Table 14.2.13 Summary of C5 Values Pharmacodynamic Population

Table 14.2.14 Summary of Plasma RA101495 Concentrations Pharmacokinetic Population

Table 14.3.1 Overall Summary of Treatment Emergent Adverse Events Safety Population

Table 14.3.2.1 Treatment Emergent Adverse Events by System Organ Class, and Preferred Term Safety Population

Table 14.3.2.2 Non-Serious Treatment Emergent Adverse Events by System Organ Class, and Preferred Term Safety Population

Table 14.3.2.3 Treatment Emergent Adverse Events by System Organ Class, Preferred Term, and Maximum Severity Safety Population

CONFIDENTAL


Review Status: Final Version: 2.0


Table 14.3.2.4 Treatment Emergent Adverse Events by System Organ Class, Preferred Term, and Relationship to Study Drug Safety Population

Table 14.3.2.5 Treatment Emergent Adverse Events Leading to Study Discontinuation by System Organ Class, and Preferred Term Safety Population

Table 14.3.2.6 Serious Treatment Emergent Adverse Events by System Organ Class, and Preferred Term Safety Population

Table 14.3.2.7 Incidence of Treatment Emergent Adverse Events by System Organ Class, Preferred Term above Reporting Frequency Threshold of 5% Safety Population

Table 14.3.2.8 Incidence of Non-Serious Treatment Emergent Adverse Events by System Organ Class, Preferred Term above Reporting Frequency Threshold of 5% Safety Population

Table 14.3.2.9 Incidence of Treatment-related Treatment Emergent Adverse Events by System Organ Class and Preferred Term Safety Population

Incidence of Treatment-related Grade 3 or greater Treatment Emergent Adverse Events by System Organ Class and Preferred Term Safety Population

Table 14.3.3.1 Thrombotic Treatment Emergent Adverse Events by System Organ Class, and Preferred Term Safety Population

Table 14.3.3.2 Hepatic Treatment Emergent Adverse Events by System Organ Class, and Preferred Term Safety Population

Table 14.3.3.3.1 Injection Site Reaction Treatment Emergent Adverse Events by System Organ Class, and Preferred Term Safety Population

Table 14.3.3.3.2 Injection Site Reactions – Details Safety Population

Table 14.3.3.4 Infection Treatment Emergent Adverse Events by System Organ Class, and Preferred Term Safety Population

Table 14.3.4.1 Summary of Clinical Chemistry Laboratory Values Safety Population

Table 14.3.4.2 Summary of Hematology Laboratory Values Safety Population

CONF

Page

CONFIDENTAL 

Review Status: Final


Table 14.3.4.3 Summary of Coagulation Laboratory Values Safety Population

Table 14.3.4.4 Summary of C-Reactive Protein and Creatine Phosphokinase Values Laboratory Values Safety Population

Table 14.3.4.5 Summary of Urinalysis Laboratory Values Safety Population

Table 14.3.4.6 Summary of Liver Function Test Values Safety Population

Table 14.3.4.8 Summary of Liver Function Test Values Safety Population

Table 14.3.4.8 Summary of PNH Clone Size Values Safety Population

Table 14.3.5 Summary of Vital Signs by Visit Safety Population

16.2.1.1 Summary of ECG Values by Visit Safety Population

16.2.1.2 Protocol Deviations Safety Population

16.2.2.1 Medical history Safety Population

16.2.2.2 PNH Disease History Safety Population

1.2.2.3 PNH Treatment history Safety Population

2.3.1 Prior Medications Safety Population

CONFIDENTAL 

Jafety Population
Listing 16.2.9.5 Pancreatic Adverse Events Safety Population
Listing 16.2.9.6 Injection Site Reaction Adverse Events Safety Population

16.2.10 Injection Ster Reactions Safety Population
2.11.1 Hematology Safety Population

...iase Safety Population
Jafety Population
Jafety Population
Jec Safety Population
Jec Safety Population
Jec Safety Population
Jec Safety Population
Jec Safety Population
Jec Safety Population
Jec Safety Population
Listing 16.2.15 Pregnancy Test Safety Population
Listing 16.2.16 Pharmacodynamic Endpoints Pharmacodynamic Population
Jec Safety Population
Jec Safety Populat

# APPENDIX II. SCHEDULE OF ASSESSMENTS

Table 1 Table Time and Events

| Analysis Plan: RA101495-01.202 APPENDIX II. SCHEI Table 1 Table Time and | DULE O | F ASS | ESSME | ENTS | | | | × 6 | in of | ereof | Review Status: Final<br>Version: 2.0<br>Version Date: 150CT2021 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| tudy Month | Screening a /Day 1a,b | 1 | 2 | 3 | 6 | 9 | 12 | Then Every<br>3 Months | Then Every<br>12 Months<br>only | Final Study<br>Visit | |
| Study Day→ | 1 | $30 \pm 7$ | 60 ± 7 | 90 ± 7 | 180 ± 7 | 270 ± 7 | 360 ± 7 | - (± 7) | - (± 7) | - | |
| Study Procedure ↓ | | | | Î | | 1 | 7 | . 0 | | | |
| Signature of ICF a | X | | | | | | | 3/0 | | | |
| Review eligibility criteria | X | | | | | X | | | | | |
| rior and Concomitant medications | X | X | X | X | X | X | X | O X | | X | |
| hysical examination | Χþ | X | X | X | X | X | X | X | | X | |
| /ital signs | ΧÞ | X | X | X | X | X | X | X | | X | |
| CG | ΧÞ | | | | | 0 | X | | X | X | |
| Blood chemistry | Хр | X | X | X | X | X | X | X | | X | |
| lematology | Хр | X | X | X | X | X | <b>x</b> | X | | X | |
| Coagulation <sup>c</sup> | Хр | X | X | X | X | X | X | X | | X | |
| Irinalysis | Хр | X | X | X | X | X | X | X | | X | |
| NH Clone size | Χp | | | X | . 🗙 | X | X | X | | X | |
| regnancy test | Хр | X | X | X | X | X | X | X | | X | |
| Quality of life assessments | Хр | X | X | X | X | X | X | X | | X | |
| dverse event monitoring (including<br>njection site reactions) | Xp | Х | Х | Х | XX | × | Х | Х | | X | |
| Pharmacokinetics <sup>d</sup> | X | X | X | X | X | X | X | | | , | |
| harmacodynamics <sup>d</sup> | X | X | X | X | X | X | X | | | | |
| Additional Biomarkers | X | X | X | X | X | X | X | | | | |
| inti-drug antibodies | X | X | X C | X | X | X | X | X | | X | |
| RA101495 dispensing and returne | X | X | X | X | X | X | X | x | | X | |
| RA101495 administration <sup>f</sup> | Xg | X | X | X | X | X | X | X | | | |

The Screening Visit should coincide with the qualifying study end of study visit and include signing of the informed consent. The informed consent should be provided to the subject prior to the qualifying study end of study visit to facilitate a proper informed consent process.

**CONFIDENTAL** 

All screening assessments are expected to be the same as those for the end of qualifying study visit and do not need to be repeated unless clinically indicated. Record AEs ongoing from qualifying All screening assessments are expected to the transfer of the study of the specific AE eCRF for ongoing AEs from the qualifying study.

Coagulation tests should be performed as per standard practice on any subject taking suficoagulant therapy in addition to specified assessments in the study.

Coagulation tests should be performed as per standard practice on any subject taking a uncoagulant merapy in addition to specified assessments PK/PD/Biomarkers sampling prior to dose on day of visit (dose held that morning and administered in clinic after blood samples are obtained). Study drug dispensing and return is monthly. Frequency of dispensing of IMP may be adjusted during the study. Study drug administration should be administered in clinic after PK and PD collection on clinic visit days for the first 12 months.